CLINICAL TRIAL: NCT03880240
Title: Gamma Induction for Amyloid Clearance in Alzheimer's Disease
Brief Title: Gamma Induction for Alzheimer's Disease
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Beth Israel Deaconess Medical Center (Other); National Institutes of Health (NIH) (NIH); National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Emiliano Santarnecchi, Associate Professor of Radiology, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2019P000092; R01AG060981 (NIH)
Record Dates: First submitted 2019-03-15; First posted 2019-03-19 (Actual); Last update posted 2023-12-06 (Actual); Status verified 2023-12

CONDITIONS: Alzheimer Disease; Mild Cognitive Impairment
Keywords: Alzheimer Disease; Mild Cognitive Impairment
MeSH Terms: conditions — Alzheimer Disease; Cognitive Dysfunction | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (4):
- 2 weeks of daily tACS sessions (Experimental): 10 daily (Monday-Friday) 1-hour sessions of tACS stimulation
  Interventions: Device: Transcranial Alternating Current Stimulation (tACS)
- 4 weeks of daily tACS sessions (Experimental): 20 daily (Monday-Friday) 1-hour sessions of tACS stimulation
  Interventions: Device: Transcranial Alternating Current Stimulation (tACS)
- 4 weeks of twice daily tACS sessions (Experimental): 20 days (Monday-Friday) of 1-hour sessions of tACS twice per day
  Interventions: Device: Transcranial Alternating Current Stimulation (tACS)
- 2/4 weeks of Sham tACS sessions (Sham Comparator): 10/20 days (Monday-Friday) of 1-hour sessions of tACS once/twice per day
  Interventions: Other: Sham Transcranial Alternating Current Stimulation

INTERVENTIONS:
Device: Transcranial Alternating Current Stimulation (tACS) — tACS is a non-invasive way of stimulating the brain externally using weak electric currents. Electrodes are placed into a cap that you wear on your head. A weak electrical current travels back and forth through the electrodes to your head. tACS will be applied at a frequency of 40Hz and targeting the area of maximal tracer uptake on amyloid PET imaging using an individualized multielectrode design to maximize the induced electrical current to the target region.
  Other Names: Non-invasive Brain Stimulation
  Arms: 2 weeks of daily tACS sessions; 4 weeks of daily tACS sessions; 4 weeks of twice daily tACS sessions
Other: Sham Transcranial Alternating Current Stimulation — Placebo Control, simulation of transcranial alternating current stimulation without receiving any stimulation
  Arms: 2/4 weeks of Sham tACS sessions

SUMMARY:
Alzheimer's Disease (AD) is characterized by amyloid-β (Aβ) plaque buildup and phosphorylated tau (p-tau) in the brain, as well as widespread neurodegeneration. Amyloid-β and tau are proteins that build up in the brain that may contribute to memory problems. The evidence suggests that both amyloid and tau play a critical role in AD and interventions that reliably and safely decrease the intracerebral burden of amyloid or tau could potentially be of marked clinical importance. Currently, therapeutic options are very limited and while there are pharmacologic interventions that transiently improve cognitive function, there are no treatments that alter disease progression.

The purpose of this study is to see if multiple daily sessions of non-invasive brain stimulation can affect brain activity to decrease the amount of amyloid and tau in people with AD as compared to Sham (placebo) stimulation. The type of brain stimulation that will be used is called transcranial alternating current stimulation (tACS). This study will investigate different doses of tACS (2-4 weeks) and assess safety. The hope is that tACS will decrease the amount of amyloid and tau and improve memory and thinking in people with AD.

DETAILED DESCRIPTION:
This is an interventional, sham controlled, double-blind study in patients with early to moderate Alzheimer's Disease (AD). The study will enroll approximately 55 individuals with amyloid positive Mild Cognitive Impairment (MCI) or AD. Each subject will undergo a 1-2 visit screening period consisting of a physical and neurological exam, medical history and medication review, safety questionnaires, and cognitive testing. Each subject will then undergo 5-7 baseline visits including neuropsychological testing (memory and thinking tests), amyloid Positron Emission Tomography (PET) imaging if one is not available or it has been greater than 6 months, tau PET imaging, tACS-EEG (transcranial alternating current stimulation and electroencephalogram) assessment, TMS-EEG (transcranial magnetic stimulation and electroencephalogram) plasticity assessment, functional magnetic resonance imaging (fMRI), blood and saliva sample collection, and optional lumbar puncture (LP). Participants will be randomly assigned to one of four groups: stimulation for 2 weeks or 4 weeks, once a day or twice a day. One of the groups is a sham group. This means that this group will not receive actual tACS. Each session will be one hour of either individualized gamma-frequency (40 Hz) tACS or sham tACS, depending on the assigned group. Subjects will be assessed for any side effects before and after each session and complete a short memory and thinking test either daily or weekly. At the end of the daily sessions, 5-7 follow up visits will include a repeat of the baseline measures including amyloid and tau PET scans. Long-term follow-up visits will include an EEG, cognitive testing and an amyloid PET scan. The PET imaging studies will be conducted at Massachusetts General Hospital and up to 5 PET scans will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Clinical Diagnosis of early to moderate AD*

  * Mini Mental State Examination (MMSE) ≥ 18
  * Clinical Dementia Rating (CDR) ≥ 0.5
  * Demonstration or history of memory impairments.

    * Confirmation of diagnosis will be made by the study MD based on a holistic consideration of the participant's cognitive evaluation and history.
* Amyloid positive PET imaging
* At least 45 years old
* On a stable dose of medications for memory loss including cholinesterase inhibitors (e.g. donepezil, rivastigmine or memantine) as defined as 6 consecutive weeks of treatment at an unchanging dose
* Minimum of completed 8th grade education
* No history of intellectual disability

Exclusion Criteria:

* Current history of poorly controlled migraines including chronic medication for migraine prevention
* Current or past history of any neurological disorder other than dementia, such as epilepsy, stroke (cortical stroke), progressive neurologic disease (e.g. multiple sclerosis) or intracranial brain lesions; and history of previous neurosurgery or head trauma that resulted in residual neurologic impairment.

  * Non-cortical disease such as confluence white matter changes (including lacunar infarcts < 1cm) and asymptomatic, subacute, cerebellar infarcts may be included upon review of a medically responsible neurologist.
* Past or current history of major depression, bipolar disorder or psychotic disorders, or any other major psychiatric condition.
* Contraindication for undergoing MRI or receiving TMS or tACS,
* >50 mSv of radiation exposure for research within the past year (PET imaging exclusion)
* History of fainting spells of unknown or undetermined etiology that might constitute seizures.
* History of seizures, diagnosis of epilepsy, history of abnormal (epileptiform) EEG or immediate (1st degree relative) family history of epilepsy; with the exception of a single seizure of benign etiology (e.g. febrile seizure) in the judgment of the investigator.
* Chronic (particularly) uncontrolled medical conditions that may cause a medical emergency in case of a provoked seizure (cardiac malformation, cardiac dysrhythmia, asthma, etc.).
* Metal implants (excluding dental fillings) or devices such as pacemaker, medication pump, nerve stimulator, TENS unit, ventriculo-peritoneal shunt, cochlear implant, unless cleared by the study MD.
* Substance abuse or dependence within the past six months.
* Medications will be reviewed by the responsible MD and a decision about inclusion will be made based on the following: The patient's past medical history, drug dose, history of recent medication changes or duration of treatment, and combination of CNS active drugs.
* All female participants that are pre-menopausal will be required to have a pregnancy test; any participant who is pregnant or breastfeeding will not be enrolled in the study.
* Subjects who, in the investigator's opinion, might not be suitable for the study
* A hair style or head dress that prevents electrode contact with the scalp or would interfere with the stimulation (for example: thick braids, hair weave, afro, wig)

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Estimated)
Dates: Start 2019-08-05 (Actual); Primary Completion 2024-11 (Estimated); Study Completion 2024-11 (Estimated)

PRIMARY OUTCOMES:
PET amyloid burden | up to 16 weeks
  Changes in the amyloid load observed via PET imaging will be evaluated by comparing PET data acquired before and after the tACS sessions
PET tau deposition | up to 16 weeks
  Changes in the tau deposition observed via PET imaging will be evaluated by comparing PET data acquired before and after the tACS sessions
Incidence of Treatment-Emergent Adverse Events | up to 16 weeks
  Adverse Events as a result of tACS stimulation will be reported
Change in Gamma activity | up to 16 weeks
  Changes in oscillatory activity in the EEG gamma band will be evaluated before and after the tACS sessions.
Alzheimer's Disease Assessment Scale -Cog Score | up to 16 weeks
  Change in ADAS-Cog score will be reported, to document a potential clinical benefit of tACS. The scale ranges from a total score of 0-70 with higher score indicating greater cognitive impairment.
  The ADAS-Cog has a total scoring range of 0-70, with the score based on the number of errors made in each of the 11 following items: word recall task, commands, constructional praxis, naming task, ideational praxis, orientation, word recognition, remembering word recognition test instructions, comprehension of spoken language, word-finding difficulty in spontaneous speech, and spoken language ability. Subscale scores are not reported, only the total score.

SECONDARY OUTCOMES:
Follow-up Amyloid PET burden | up to 16 weeks
  Changes in the amyloid load observed via PET imaging at follow-up visits.
Follow-up Cognitive Evaluation | up to 16 weeks
  Changes in Alzheimer's Disease Assessment Scale-Cognitive (ADAS-Cog) score at follow-up visits
  The ADAS-Cog has a total scoring range of 0-70, with the score based on the number of errors made in each of the 11 following items: word recall task, commands, constructional praxis, naming task, ideational praxis, orientation, word recognition, remembering word recognition test instructions, comprehension of spoken language, word-finding difficulty in spontaneous speech, and spoken language ability. Subscale scores are not reported, only the total score.
  The scale ranges from a total score of 0-70 with higher score indicating greater cognitive impairment.

CONTACTS AND LOCATIONS:
Overall Officials: Emiliano Santarnecchi, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States